CLINICAL TRIAL: NCT05422664
Title: A Multicenter Clinical Study of Acute Sympotomatic Seizure Secondary to Autoimmune Encephalitis and Autoimmune-associated Epilepsy
Brief Title: Acute Sympotomatic Seizure Secondary to Autoimmune Encephalitis and Autoimmune-associated Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Liu Yonghong (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Xian Children's Hospital (Other Government); Baoji Central Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Qilu Children's Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Liu Yonghong, professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: KY20222079-F-1
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Autoimmune Encephalitis; Epilepsy; Seizures
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Lacosamide — Patients with autoimmune related epilepsy were included. After obtaining informed consent, lacosamide was given according to the weight of the patients, and the efficacy and safety were observed.

SUMMARY:
Previously, scholars called the seizures secondary to autoimmune encephalitis（AE） "autoimmune related epilepsy", but the seizures secondary to AE are usually controlled after the improvement of encephalitis, which does not meet the "persistent" characteristics of epilepsy. Only a subset of patients with seizures lasting several years require long-term Antiseizure medications (ASM). In 2020, the International Coalition against Epilepsy classified it as "acute symptomatic seizure secondary to AE". ASSAE) and autoimmune-associated epilepsy (AAE) . The former is caused by AE, which has clinical manifestations of AE at the same time as epileptic seizures at the beginning or recurrence. The proportion and type of epileptic seizures are different due to different causes, and epileptic seizures are also controlled after the disease is controlled. The latter is that after adequate immunotherapy, there are still persistent seizures, and there is no obvious evidence of inflammatory activity, this type of patient application ASM and immunotherapy is not effective.

Secondly, with the deepening of AE research, gradually found that some AAE can still be ASMs cure, such as carbamazepine, ocasepine, lakaosamine. On the one hand, it works by influencing cellular and humoral immune responses. On the other hand, effectiveness of sodium channel blockers in focal epilepsy. Lacosamide is a slow sodium channel blocker that belongs to the third generation of ASM. It has a short half-life and can be quickly increased to an effective dose with a low incidence of adverse reactions. Therefore, the investigators chose to add oral antiepileptic therapy with lacosamide in AAE populations to observe efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed autoimmune encephalitis (2016,Lancet);
2. Meet the classification criteria for epilepsy (2017,International League Against Epilepsy);
3. Patients who still have seizures after taking ASM after the control of AE disease were included in the third part of the study;
4. All patients volunteered and signed an informed consent form;

Exclusion Criteria:

1. Incomplete key clinical data;
2. People with epilepsy or other intracranial diseases before diagnosis;
3. There is no epileptic author during the onset of autoimmune encephalitis;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed autoimmune encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
seizures or epilepsy | From admission to discharge, up to 5 years
  Patients with autoimmune encephalitis have sympotmatic seizures in the acute phase,which develop into seizure-free or autoimmune-associated epilepsy.
seizure-free or others | 1 year after lacosamide addition
  After obtaining informed consent, patients who eventually developed autoimmune epilepsy were given oral antiepileptic therapy with lacosamide according to their body weight, and the remission of seizures was observed.

CONTACTS AND LOCATIONS:
Locations (1):
- XijingH, Xi'an, Shaanxi, China